CLINICAL TRIAL: NCT00743067
Title: A Phase 1 Dose Escalation Study of the Safety and Pharmacokinetics of GSK1363089 (Formerly XL880) Administered Orally Daily to Subjects With Solid Tumors
Brief Title: A Dose Escalation Study of the Safety and Pharmacokinetics of GSK1363089 (Formerly XL880) Administered Orally Daily to Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MET111648; NCT00349609 (obsolete NCT alias)
Record Dates: First submitted 2008-08-26; First posted 2008-08-28 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Solid Tumours
Keywords: XL880; MET inhibitor; GSK1363089; Solid Tumors; c-Met
MeSH Terms: interventions — GSK 1363089

ARMS (5):
- Cohort 1 (Experimental): Cohort 1 will include 60 milligram (mg) of GSK1363089. Dose escalation will be 100% if there is no drug-related AEs of Grade 2 or higher in previous cohort. Dose escalation will be 50% in case there is Grade 2 drug-related AEs in any previous cohort.
  Interventions: Drug: GSK1363089 (formerly XL880)
- Cohort 2 (Experimental): Cohort 2 will include 120 mg of GSK1363089. Dose escalation will be 100% if there is no drug-related AEs of Grade 2 or higher in previous cohort. Dose escalation will be 50% in case there is Grade 2 drug-related AEs in any previous cohort.
  Interventions: Drug: GSK1363089 (formerly XL880)
- Cohort 3 (Experimental): Cohort 3 will include 240 mg of GSK1363089. Dose escalation will be 100% if there is no drug-related AEs of Grade 2 or higher in previous cohort. Dose escalation will be 50% in case there is Grade 2 drug-related AEs in any previous cohort.
  Interventions: Drug: GSK1363089 (formerly XL880)
- Cohort 4 (Experimental): Cohort 4 will include 480 mg of GSK1363089. Dose escalation will be 100% if there is no drug-related AEs of Grade 2 or higher in previous cohort. Dose escalation will be 50% in case there is Grade 2 drug-related AEs in any previous cohort.
  Interventions: Drug: GSK1363089 (formerly XL880)
- Cohort 5 (Experimental): Cohort 5 will include 960 mg of GSK1363089. Dose escalation will be 100% if there is no drug-related AEs of Grade 2 or higher in previous cohort. Dose escalation will be 50% in case there is Grade 2 drug-related AEs in any previous cohort.
  Interventions: Drug: GSK1363089 (formerly XL880)

INTERVENTIONS:
Drug: GSK1363089 (formerly XL880) — GSK1363089 will be available as solid capsules with dose unit of 20, 100 and 200 mg. Subjects will administer GSK1363089 capsules orally

SUMMARY:
This clinical study is being conducted at two sites to determine the optimum dose, safety, and tolerability of oral daily GSK1363089 treatment in adults with solid tumors. This study is no longer recruiting subjects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor which is metastatic or unresectable with no known effective treatment measures,
* ECOG performance status of </= 2.
* Adequate bone marrow reserve, hepatic, renal, and cardiovascular function,
* Negative pregnancy test.

Exclusion Criteria:

* Anticancer therapy within 30 days of the start of treatment,
* Received radiation to =25% of bone marrow within 30 days of treatment.
* Known brain metastasis,
* Uncontrolled intercurrent illness,
* HIV positive,
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2006-08-09 (Actual); Primary Completion 2009-05-02 (Actual); Study Completion 2009-11-09 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) and to evaluate the safety and tolerability of daily oral administration of GSK1363089 in subjects with solid tumors | 2 years

SECONDARY OUTCOMES:
Plasma pharmacokinetics (PK) of daily GSK1363089 in subjects with solid tumors, pharmacodynamic effects of daily GSK1363089, Long-term safety and tolerability of daily GSK1363089, Tumor response after daily administration of GSK1363089 | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Shapiro GI, McCallum S, Adams LM, Sherman L, Weller S, Swann S, Keer H, Miles D, Muller T, Lorusso P. A Phase 1 dose-escalation study of the safety and pharmacokinetics of once-daily oral foretinib, a multi-kinase inhibitor, in patients with solid tumors. Invest New Drugs. 2013 Jun;31(3):742-50. doi: 10.1007/s10637-012-9881-z. Epub 2012 Oct 6. PMID 23054208
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study MET111648 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/MET111648?search=study&search_terms=MET111648#rs
- Available data/document: Dataset Specification: MET111648 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: MET111648 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: MET111648 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: MET111648 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: MET111648 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: MET111648 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: MET111648 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register